CLINICAL TRIAL: NCT02677688
Title: Restauration of EBV Control in SLE Phase 1-2 Trial Evaluating Adoptive Transfer of Autologous EBV- Specific Cytotoxic T Lymphocytes in SLE Treatment
Brief Title: Autologous EBV-specific Cytotoxic T Cells for the Treatment of Systemic Lupus Erythematosus (SLE)
Acronym: LUPUS CTL EBV
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: completed inclusions
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/10/06-X
Record Dates: First submitted 2016-01-28; First posted 2016-02-09 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Serologically Active Adult Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; autologous anti-EBV CTL; adoptive therapy; phase 1 -2
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous EBV specific CTL infusion (Experimental)
  Interventions: Biological: Autologous EBV specific CTL infusion

INTERVENTIONS:
Biological: Autologous EBV specific CTL infusion

SUMMARY:
EBV has been implicated in pathogeny of SLE with increase in EBV sero-prevalence, defective control in EBV infection and altered both B and T immune responses to this virus The main objective of this pilot proof-of-concept (POC) study is to evaluate safety and efficacy of autologous EBV specific CTL adoptive transfer in adult patients with serologically active SLE

DETAILED DESCRIPTION:
Systemic lupus is a disabling disease of the young woman, whose treatment is based on the long-term corticosteroid, anti-malarials and immunosuppressants synthesis. This support is not without potential side effects. EBV is a herpes causes infectious mononucleosis virus, usually encounter in childhood or adolescence, and that our natural immunity cell (CD8 T cells) controls all our lives, not eliminate.

Increasingly scientific studies show that there are patients with systemic lupus (and multiple sclerosis), a failure of self-control of the EBV virus, by T lymphocytes (CD8). This uncontrolled virus then stimulate the B lymphocytes, which produce antibodies, toxic in lupus. The laboratory isolate T cells specific for EBV (EBV-CTL) of a patient, and stimulate in culture to strengthen them. They can be then re-injected by a single intravenous infusion (autotransfusion), and were used to control the virus in certain diseases where EBV has a demonstrated role post-transplant lymphoproliferative disorder, chronic fatigue syndrome EBV-induced.

Our therapeutic approach is completely innovative, as based on the principle of cell therapy, thus not using new drugs, and based on the restoration of the patient's immune system, specific EBV.

ELIGIBILITY:
Inclusion Criteria:

* 4 systemic lupus criteria of the American College of Rheumatology with antinuclear antibodies> 1:80
* Age greater than or equal to 18 years
* Lupus serologically active without active serious disease (Kidney, CNS)
* Anti-native DNA Ac positive and / or C3 or C4 low
* SLEDAI greater than or equal to 2 at baseline
* Serology HBV, HCV, HIV, HTLV-1, syphilis: Negative J-30 before sample
* Hemoglobin >11g/dL
* Prednisone dose <15 mg / day with a stable dose within 30 days previous injection
* Immunosuppressive treatments which dosage has not been increased for at least 3 months before enrollment
* Agreement telephone and / or mail for coordinating investigator inclusion
* Social ensured Patient
* EBV positive serology

Exclusion Criteria:

* Evolving severe lupus, requiring high dose corticosteroids and / or immunosuppressive therapy
* Psychiatric disorders
* Predicted Failure to monitoring compliance with impossibility
* Infectious Episode underway
* Evolutionary Cancer
* Risk of death within 6 months
* Consent Refusal
* Pregnancy
* Nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
description of adverse events according CTC toxicity criteria . | month 12
  Tolerance will be assessed by clinical and laboratory examinations to each Visit according to CTC toxicity criteria.

SECONDARY OUTCOMES:
Systemic Lupus Erythematosus clinical activity | day 0, day 10, week 4, month 3, month 6, month 9 and month 12
  Composite Response of SLE Index (Systemic Lupus Erythematosus Responder Index: Systemic Lupus Erythematosus Disease Activity Index + British Isles Lupus Assessment Group + Physician Global Assessment)
Quality of Life, The Short Form (36) Health Survey | day 0, day 10, week 4, month 3, month 6, month 9 and month 12
  The Short Form (36) Health Survey
Lupus Quality of Life | day 0, day 10, week 4, month 3, month 6, month 9 and month 12
  Lupus Quality of Life questionnaire
Systemic Lupus Erythematosus biological activity (1) | day 0, day 10, week 4, month 3, month 6, month 9 and month 12
  biological parameter measurement biomarkers C3
Systemic Lupus Erythematosus biological activity (2) | day 0, day 10, week 4, month 3, month 6, month 9 and month 12
  biological parameter measurement biomarkers C4
Systemic Lupus Erythematosus biological activity (3) | day 0, day 10, week 4, month 3, month 6, month 9 and month 12
  biological parameter measurement biomarkers anti-dsDNA antibodies
Systemic Lupus Erythematosus biological activity (4) | day 0, day 10, week 4, month 3, month 6, month 9 and month 12
  biological parameter EBV blood load

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamidou, PU PH, Study Director — Nantes University Hospital
Locations (3):
- France (3):
  - CHU de Nantes - Dermatologie, Nantes
  - CHU de Nantes - Médecine interne, Nantes
  - Hopital La pitié Salpétriere, Paris

IPD SHARING:
Plan to Share IPD: No